CLINICAL TRIAL: NCT06886633
Title: The Effect of Breathing Exercise and Pressurized Cold Application on Pain and Anxiety During Sharp Debridement in Diabetic Foot Ulcers
Brief Title: The Effect of Breathing Exercise and Pressurized Cold Application on Pain and Anxiety During Sharp Debridement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma Aslan, Nurse, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Hasan Kalyoncu University
Record Dates: First submitted 2024-12-23; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Debridement; pain; anxiety; Breathing Exercise; Pressurized Cold Application
MeSH Terms: conditions — Diabetic Foot; Pain; Anxiety Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Breathing Exercise Group (Experimental): Volunteering to participate in the study, Being 18 years of age or older, Not having a disease that affects breathing such as asthma, COPD, heart failure, Not taking any medication that suppresses anxiety symptoms, Not having a disease that prevents communication such as Alzheimer's or dementia, Not having problems with the ear, nose or throat,
  Interventions: Behavioral: Breathing exercise
- Pressurized Cold Application Group (Experimental): Volunteering to participate in the study, Being 18 years of age or older, Not having a disease that affects breathing such as asthma, COPD, heart failure, Not taking any medication that suppresses anxiety symptoms, Not having a disease that prevents communication such as Alzheimer's or dementia, Not having problems with the ear, nose or throat,
  Interventions: Device: Experimental: Pressurized Cold Application Group
- control group (No Intervention): Volunteering to participate in the study, Being 18 years of age or older, Not having a disease that affects breathing such as asthma, COPD, heart failure, Not taking any medication that suppresses anxiety symptoms, Not having a disease that prevents communication such as Alzheimer's or dementia, Not having problems with the ear, nose or throat,

INTERVENTIONS:
Behavioral: Breathing exercise — Patients participating in the breathing exercise group will be trained to apply the breathing exercise at least 1 hour before starting the debridement process. 5 minutes before starting the debridement procedure, the researcher will start breathing exercises in the patient's room. The exercise duration will be approximately 15-20 minutes, and the environment will be quiet, at room temperature and well ventilated during the exercise.
  The gel part of the pressurized cold therapy bandage will be removed and kept in the refrigerator for at least 2 hours to make it ready for application. The cold gel pack removed from the freezer section of the refrigerator will be placed inside the pressurized cold therapy bandage before application. Pressurized cold will be applied to the patient 10 minutes before starting the debridement procedure.
  Arms: Breathing Exercise Group
Device: Experimental: Pressurized Cold Application Group — The gel part of the pressure cold therapy bandage will be removed and kept in the refrigerator for at least 2 hours to make it ready for application, and the cold gel pack taken from the freezer section of the refrigerator before application will be placed inside the pressure cold therapy bandage. Pressure cold will be applied to the patient 10 minutes before starting the debridement procedure. The patient will be assessed and recorded by a nurse independent of the research on the State Anxiety Scale before and after debridement, and the Visual Comparison Scale before, during and after debridement.
  Arms: Pressurized Cold Application Group

SUMMARY:
In our planned study, it is envisaged that patients who receive breathing exercises and pressurized cold application will experience a decrease in the level of pain they feel during the debridement process, a decrease in their anxiety levels, and an improvement in their vital signs, and that these study findings will constitute an important data source to reduce the pain and anxiety that occurs during the debridement process.

DETAILED DESCRIPTION:
Approximately half of the diabetic population is at risk for developing foot ulcers. A prevalence study conducted in our country stated that more than 1 million of 7 million patients with diabetes developed diabetic foot ulcers (DAU) and nearly 500,000 patients had diabetic foot infections. Diabetic foot ulcers cause deterioration in the patient's quality of life, significant increase in treatment costs, lower extremity amputations and increased mortality. 50-70% of non-traumatic foot amputations are performed on diabetic foot patients .

When the literature is examined, it is seen that breathing exercises have been used to support the treatment of stress, fatigue and pain since human history. Breathing exercise is a method that ensures body-mind harmony. Conscious deep and slow breathing helps develop conscious control over relaxation and increases awareness. The distracting effect of breathing can be effective in relieving pain through many different mechanisms: Breathing exercises can relieve tension and muscle spasms in the body by reducing stress. Pain is often associated with stress, tension and anxiety. The rhythmic and regular movement of breathing can help calm the mind and become less sensitive to pain. It may increase the release of natural painkillers called endorphins. Deep breathing and relaxation can trigger the release of endorphins in the brain and reduce the perception of pain. There are studies that breathing exercise increases the pain threshold, reduces the level of anxiety by allowing the person to relax, and has healing effects on vital signs.

Cold application is used as an effective alternative treatment to relieve pain and is recommended because it reduces pain as a result of its effect on sensory nociceptors. Compression increases conductivity by ensuring full contact between ice and skin, and reduces blood flow and edema to the tissue by strengthening the effect of cold application in reducing tissue temperature. For this reason, it is stated that using cold and pressure together is a more effective method to reduce the level of pain than applying cold alone. It has been reported that pressurized cold application is an important application in reducing the level of pain in patients undergoing total knee prosthesis. There are studies showing that cold application reduces both the level of pain and the level of anxiety.

It has been reported that cold saline application and stress ball application to reduce pain and anxiety during wound debridement in patients with diabetic foot ulcers reduce the level of pain and anxiety during debridement. According to the literature, there are limited studies on reducing pain and anxiety during debridement in diabetic foot ulcer patients. In our planned study, it is envisaged that patients who receive breathing exercises and pressurized cold application will experience a decrease in the level of pain they feel during the debridement process, a decrease in their anxiety levels, and an improvement in their vital signs, and that these study findings will constitute an important data source to reduce the pain and anxiety that occurs during the debridement process. At the same time, it is thought that using it as an alternative to the use of medication to reduce the level of pain during the procedure will make a significant contribution to reducing treatment costs.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Those aged 18 and over,
* Those who were included in the breathing exercise group before the research and who could perform breathing exercises correctly if taught and demonstrated.
* Do not have a disease that affects breathing such as Asthma, COPD, Heart failure,
* Not taking any medication that suppresses anxiety symptoms,
* Do not have a diagnosed disease such as Alzheimer's or Dementia that would hinder communication,
* Patients included in the breathing exercise group should not have ear, nose or throat problems that may prevent them from performing breathing exercises.

Exclusion Criteria:

* Those who give up being a research participant at any stage of the research,
* Illiterate
* Having a diagnosed disease that affects breathing such as Asthma, COPD, Heart failure,
* Taking any medication that suppresses anxiety symptoms,
* Cold intolerance or allergy to cold

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Scale | Breathing exercises will be performed 5 minutes before starting the debridement process. The exercise will last approximately 15-20 minutes, and the State Anxiety Scale will be administered before and 5 minutes after debridement process.
  The State Anxiety Inventory (STAI-I) was developed by Spielberger in 1970, adapted to Turkish by Öner N et al. and its validity and reliability study was conducted. The anxiety level is scored as "(1) not at all, (2) a little, (3) a lot and (4) completely" in the STAI-I. Items 3, 4, 6, 7, 9, 12, 13, 14, 17, and 18 in the inventory are positive for 40 (increase total anxiety), and items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 are positive (decrease total score). The total score of the reverse statements is subtracted from the total score obtained for direct statements. In scoring, a score between 1 (or -1) and 4 (or -4) is expected for each item according to its positive or negative feature, and 50 is added to the total score to be obtained. The highest score is 80, the lowest score is 20. The higher the total anxiety score, the more anxiety the person has.
Visual Analog Scale | The patient will be applied compressive cold 10 minutes before the debridement process. A visual comparison scale will be applied to the patient before, during and 5 minutes after debridement process
  The Turkish validity and reliability of this scale, which was developed by Price et al. (1994) to assess the severity of pain, was conducted by Eti Aslan (2004) by assessing the presence of pain in patients in the postoperative period. The scale is graded from 0 to 10, with 0 = no pain, and 10 = unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Background] Chen CT, Tung HH, Chen YC, Wang JL, Tsai SH, Huang YT, Hsu TF. Cold application for pain and anxiety reduction following chest tube removal: A systematic review and meta-analysis. J Clin Nurs. 2023 Feb;32(3-4):574-583. doi: 10.1111/jocn.16315. Epub 2022 Apr 6. PMID 35388557
- [Background] Hu L, Hua Y, Wang L, Mao Z, Jia X, Lei Z, Chang D, Cheng W. Effect of Short-term Deep Breathing Exercises on Perioperative Anxiety and Pain in Pediatric Orthopedic Patients: A Randomized Controlled Trial. J Perianesth Nurs. 2025 Feb;40(1):69-75. doi: 10.1016/j.jopan.2024.03.009. Epub 2024 Jul 9. PMID 38980240
- [Background] Dayya D, O'Neill OJ, Huedo-Medina TB, Habib N, Moore J, Iyer K. Debridement of Diabetic Foot Ulcers. Adv Wound Care (New Rochelle). 2022 Dec;11(12):666-686. doi: 10.1089/wound.2021.0016. Epub 2021 Dec 21. PMID 34376065